CLINICAL TRIAL: NCT02243319
Title: A Randomized, Open Label, Crossover Study to Investigate the Pharmacokinetic Drug Interactions Between HGP1201 and HGP0904 in Healthy Male Subjects
Brief Title: Investigating the Pharmacokinetic Drug Interactions Between HGP1201 and HGP0904
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-TARO-101
Record Dates: First submitted 2014-08-24; First posted 2014-09-17 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): A → B → C
  A: HGP1201 for 9 days B: HGP0904 for 9 days C: HGP1201+ HGP0904 for 9 days
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion
- Group 2 (Experimental): C → A → B
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion
- Group 3 (Experimental): B → C → A
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion
- Group 4 (Experimental): C → B → A
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion
- Group 5 (Experimental): B → A → C
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion
- Group 6 (Experimental): A → C → B
  Interventions: Drug: HGP1201; Drug: HGP0904; Drug: HGP0904 and HGP1201 co-administraion

INTERVENTIONS:
Drug: HGP1201
Drug: HGP0904
Drug: HGP0904 and HGP1201 co-administraion

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic drug interactions between HGP1201 and HGP0904

DETAILED DESCRIPTION:
Randomized, open-label, multiple dose , 3-treatment, 6-sequence, 3-period, crossover study, The purpose of this study is to investigate the pharmacokinetic drug interactions between HGP1201 and HGP0904

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer, age 19~45 years
* The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 28 kg/m2
* Subject who has the ability to comprehend the study objectives, contents and the property of the study drug before participating in the trial.

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study
* History of relevant drug allergies or clinically significant hypersensitivity reaction.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of HGP1201, HGP0904 | 1D 0h(predose), 8D 0h, 9D 0h, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 10D 0h, 11D 0h, 12D 0h
AUCτ,ss of HGP1201, HGP0904 | 1D 0h(predose), 8D 0h, 9D 0h, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 10D 0h, 11D 0h, 12D 0h

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Seok Lim, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No